CLINICAL TRIAL: NCT01234909
Title: The Atopic Dermatitis Clinic as an Entry Point for Community Outreach in Asthma, Missed Immunizations, and Vitamin D Deficiency
Brief Title: Asthma, Missed Immunizations, and Vitamin D Deficiency in Atopic Dermatitis
Status: Terminated | Type: Observational
Why Stopped: Not meeting enrollment goals.
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Children's Hospital and Health System Foundation, Wisconsin (Other)
Responsible Party: Principal Investigator, Yvonne Chiu, Assistant Professor, Medical College of Wisconsin
Other Study IDs: CHW 10/129, GC 1141
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Atopic Dermatitis; Vitamin D Deficiency; Asthma
Keywords: Missed immunizations
MeSH Terms: conditions — Dermatitis, Atopic; Vitamin D Deficiency; Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Atopic dermatitis: Pediatric patients ages 1-18 years old with atopic dermatitis

SUMMARY:
Atopic dermatitis is a chronic skin disease with pruritus as one of its main features. Because of the symptomatic nature of their condition, pediatric patients with atopic dermatitis may preferentially seek care in the subspecialty dermatology clinic while falling behind in visits to their primary care provider. This cross-sectional study in patients attending the Dermatology Clinic at Children's Hospital of Wisconsin will screen for common conditions associated with atopic dermatitis and subsequently treat or refer patients for appropriate care. The investigators hypothesize that Milwaukee County pediatric patients with atopic dermatitis will have a high prevalence of asthma needing treatment, missed immunizations requiring catch-up, and vitamin D deficiency necessitating replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with atopic dermatitis by a Children's Hospital of Wisconsin (CHW) pediatric dermatologist
* Age 1- 18 years old
* Primary residence in Milwaukee County

Exclusion Criteria:

* Other chronic, systemic diseases other than asthma or environmental allergies
* Hyperimmunoglobulin E or Job syndrome
* Ichthyosis disorder other than ichthyosis vulgaris
* Prior systemic therapy or phototherapy for atopic dermatitis
* Ongoing or prior treatment for known Vitamin D deficiency
* On chronic systemic corticosteroids for asthma

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children's Hospital of Wisconsin Pediatric Dermatology clinic
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Chiu, MD, Principal Investigator — Children's Hospital and Health System Foundation, Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States